CLINICAL TRIAL: NCT02751255
Title: A Phase 1 and Phase 2 Study of Daratumumab in Combination With All-trans Retinoic Acid in Relapsed/Refractory Multiple Myeloma
Brief Title: Daratumumab in Combination With ATRA
Acronym: DARA/ATRA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Erasmus Medical Center (Other); UMC Utrecht (Other); University of Turin, Italy (Other); Vejle Hospital (Other)
Responsible Party: Principal Investigator, WCJ van de Donk, Hematologist, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-003862-10
Record Dates: First submitted 2016-04-04; First posted 2016-04-26 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- daratumumab--> daratumumab + ATRA (Experimental): In part A of the study patients will be treated with daratumumab as a single agent. In case patients have progressive disease after cycle 1, or in case patients achieve less than minimal response after cycle 2, or patients achieve less than PR after cycle 3, or in case patients experience progression during daratumumab therapy after having obtained a response, then ATRA will be added to daratumumab (part B).
  Interventions: Drug: all-trans retinoic acid (ATRA)

INTERVENTIONS:
Drug: all-trans retinoic acid (ATRA) — Phase 1 and 2: daratumumab 16 mg/kg, first 8 infusions are given weekly, then 8 infusions every 3 weeks, then every 4 weeks until progression Phase 1: ATRA 15, 30, or 45 mg/m2/day for 3 days. Phase 2: ATRA will be administered twice daily as an oral formulation at the MTD dose, or if no MTD is reached, at the dose of 45 mg/m2/day for 3 days. The first administration of ATRA will be given in the morning, two days before the scheduled daratumumab infusion. The last administration of ATRA will be given in the evening of the day that daratumumab was administered (days -2, -1, and 0; day 0 is the day of daratumumab infusion).
  Other Names: ATRA

SUMMARY:
Multiple myeloma (MM) patients who develop bortezomib and lenalidomide-resistant disease have a very poor survival of only a median of 9 months, indicating that new agents are urgently needed. Recent studies have shown that daratumumab as a single agent is effective and well tolerated in these heavily pretreated MM patients. However, approximately 60% of patients do not achieve a partial response, and ultimately all patients will develop progressive disease during daratumumab therapy.

The investigators have demonstrated that levels of the target antigen CD38, and expression levels of the complement inhibitory proteins CD55 and CD59 determine the susceptibility of the MM cells towards daratumumab. In addition, MM cells have lower CD38 expression levels and higher levels of CD55/CD59 at the time of progression. Importantly, all-trans retinoic acid (ATRA) upregulates CD38 levels and downregulates CD55/CD59 levels on MM cells, both in daratumumab naïve cells and in cells that are resistant to daratumumab because of previous exposure to this drug. These alterations in expression explain the strong synergy between ATRA and daratumumab, both in MM cells derived from daratumumab naïve patients and from patients with daratumumab-refractory disease.

These data form the preclinical rationale for clinical evaluation of ATRA and daratumumab in MM patients.

DETAILED DESCRIPTION:
Multiple myeloma (MM) patients that develop bortezomib and lenalidomide-resistant disease have a very poor survival of only a median of 9 months. This clearly illustrates that new anti-MM agents are needed with different mechanisms of action.

Importantly, daratumumab monotherapy is effective and well tolerated in heavily pre-treated lenalidomide and bortezomib-refractory myeloma patients. However, approximately 60% of patients do not achieve a partial response, and ultimately all patients, also those achieving complete response, will develop progressive disease during daratumumab therapy. Factors that determine the susceptibility of MM cells to daratumumab include levels of the target antigen CD38, and expression levels of the complement inhibitory proteins CD55 and CD59. At the time of progression, there is a reduced level of CD38 on the MM cells, whereas CD55 and CD59 levels are increased. This indicates that these factors are also involved in the development of daratumumab-resistant disease.

Importantly, ATRA upregulates CD38 levels and downregulates CD55/CD59 levels on MM cells, both in daratumumab naïve cells and in cells that are resistant to daratumumab because of previous exposure to this drug. These alterations in expression explain the strong synergy between ATRA and daratumumab, both in MM cells derived from daratumumab naïve patients and from patients with daratumumab-refractory disease.

These data form the preclinical rationale for clinical evaluation of ATRA and daratumumab in MM patients. The investigators will treat relapsed/refractory MM patients in two stages. The first stage (part A) consists of treatment with daratumumab monotherapy. In case these patients have progressive disease after cycle 1, less than minimal response after cycle 2, or less than partial response after cycle 3 (unless ongoing response) to single agent daratumumab, or in case these patients progress during daratumumab therapy after previous response, then ATRA will be added to daratumumab (part B).

The aims of this study are to develop a safe ATRA and daratumumab combination suitable for clinical use and evaluation in subsequent randomized clinical trials. To this end, the maximum tolerated dose (MTD) of ATRA and daratumumab will be determined for patients with relapsed/refractory disease, who were treated with daratumumab but failed to achieve a partial response, or developed progressive disease during daratumumab treatment. This will be followed by a second part in which the investigators will examine the effectivity and toxicity profile of the combination at the MTD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Subject must have documented multiple myeloma as defined by the criteria below:

   * Monoclonal plasma cells in the bone marrow ≥10% at some point in their disease history or presence of a biopsy proven plasmacytoma.
   * Measurable disease as defined by any of the following:

   Serum monoclonal paraprotein (M-protein) level ≥5 g/L (0.5 g/dL); or urine M-protein level ≥200 mg/24 hours; or serum immunoglobulin free light chain ≥100 mg/L (10 mg/dL) and abnormal serum immunoglobulin kappa lambda free light chain ratio (See Appendix A)
3. Relapsed from or refractory to 2 or more different prior therapies, including immunomodulatory drugs (IMiDs; eg, thalidomide, lenalidomide) and proteasome inhibitors, chemotherapy-based regimens, or autologous stem cell transplantation (ASCT).

   * Relapse is defined as progression of disease after an initial response (MR or better) to previous treatment, more than 60 days after cessation of treatment
   * Refractory disease is defined as <25% reduction in M-protein or progression of disease during treatment or within 60 days after cessation of treatment
4. WHO performance 0, 1, or 2
5. Life expectancy at least 3 months
6. Written informed consent

Exclusion Criteria:

1. Subject has received daratumumab or other anti-CD38 therapies, within 6 months before start of treatment (however, patients treated with daratumumab monotherapy in compassionate use program or after European Medicines Agency (EMA) approval, and have progressive disease during daratumumab after previous response, or unresponsive disease to daratumumab [progressive disease after cycle 1, less than minimal response after cycle 2, or less than partial response after cycle 3], may be included in Part B)
2. Non-secretory myeloma
3. Systemic amyloid light-chain (AL) amyloidosis or plasma cell leukemia (>2.0x109/L circulating plasma cells by standard differential) or Waldenstrom's macroglobulinemia
4. Subject has known meningeal involvement of multiple myeloma
5. Subject has received anti-myeloma treatment within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, before start of treatment. This included subjects who have received a cumulative dose of corticosteroid greater than or equal to the equivalence of 140 mg prednisone or a single dose of corticosteroid greater than or equal to the equivalence of 40 mg/day dexamethasone within the 2-week period before start of treatment.
6. Subject has previously received an allogeneic stem cell transplantation within 1 year before the date of registration and has not used immunosuppressive drugs within one months before the date of registration.
7. Inadequate marrow reserve as defined by a platelet count <30 x 109/L or an absolute neutrophil count <1.0 x 109/L
8. a) Subject has known chronic obstructive pulmonary disease (COPD) with an Forced Expiratory Volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for patients suspected of having COPD and subjects must be excluded if FEV1 <50% of predicted normal.

   b) Subject has known moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification. (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study).
9. Subject has clinically significant cardiac disease, including:

   * Myocardial infarction within 6 months before Cycle 1, Day 1, or unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association Class III-IV)
   * Cardiac arrhythmia (Common Terminology Criteria for Adverse Events [CTCAE] Version 4 Grade 2 or higher) or clinically significant ECG abnormalities.
   * Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec.
10. Significant hepatic dysfunction (total bilirubin 3 times normal value or transaminases 3 times normal value), unless related to myeloma
11. Creatinine clearance <20 ml/min.
12. Known hypersensitivity to components of the investigational product or severe allergic or anaphylactic reactions to humanized products.
13. Subject has any concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, etc.) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
14. Subject is known to be seropositive for human immunodeficiency virus (HIV) or have active hepatitis B or hepatitis C.
15. History of active malignancy during the past 5 years, except squamous cell and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the local investigator, with concurrence with the principal investigator, is considered cured with minimal risk of recurrence within 5 years.
16. Subject is known or suspected of not being able to comply with the study protocol (eg, because of alcoholism, drug dependency, or psychological disorder) or the subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments.
17. Pregnant or lactating females
18. Women of childbearing potential not willing to use adequate contraception, defined as hormonal birth control or intrauterine device, during the trial and for 1 year after the last dose of daratumumab. For patients in the US, the use of a double-barrier method is also considered adequate.
19. Sensory or motor neuropathy of ≥grade 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
MTD | phase 1, during the first treatment cycle (28 days)
  To determine the maximum tolerated dose (MTD) of daratumumab combined with ATRA. MTD is defined during the first treatment cycle (4 weeks).
overall response rate | Phase 2, every 28 days, until last treatment received, estimated to be 8 months
  To investigate the efficacy of daratumumab combined with ATRA at the RDL, as determined by the overall response rate. This will be determined through study completion.
RDL | phase 1, during the first treatment cycle (28 days)
  To determine the recommended phase 2 dose level (RDL) of daratumumab combined with ATRA. RDL is defined during the first treatment cycle (4 weeks).

SECONDARY OUTCOMES:
Incidence of severe adverse events | Phase 1 and 2, throughout treatment, estimated to be 8 months
  evaluation of severe adverse events (SAEs) through study completion. The analysis of treatment toxicity will be done primarily by tabulation of the incidence of adverse events CTCAE grade 2 or more by treatment cycle. Data from all subjects who receive any study drug will be included in the safety analyses. In the by-subject analysis, a subject having the same event more than once will be counted only once. Adverse events will be summarized by worst CTCAE grade.
Progression-free survival (PFS) | phase 2, all patients will be followed until 1 year after the last patient has received the last infusion of daratumumab.
  Progression-free survival is defined as time from registration until progression or death, whichever comes first. Actuarial survival curves for PFS will be computed using the Kaplan-Meier method, and 95% confidence interval (CI) will be constructed.
overall survival (OS) | phase 2, all patients will be followed until 1 year after the last patient has received the last infusion of daratumumab.
  OS will be determined until study completion
prognostic factors for response | phase 1 and 2, every 28 days, until last treatment received, estimated to be 8 months
  This includes beta2 microglobulin (mg/L), cytogenetic abnormalities as determined by fluorescence in situ hybridization (FISH), thrombocyte counts, albumin, and LDH. These prognostic factors will be determined at baseline, before the first daratumumab infusion.
prognostic factors for PFS | phase 1 and 2, all patients will be followed until 1 year after the last patient has received the last infusion of daratumumab.
  This includes beta2 microglobulin (mg/L), cytogenetic abnormalities as determined by fluorescence in situ hybridization (FISH), thrombocyte counts, albumin, and LDH. These prognostic factors will be determined at baseline, before the first daratumumab infusion.
prognostic factors for OS | phase 1 and 2, all patients will be followed until 1 year after the last patient has received the last infusion of daratumumab.
  This includes beta2 microglobulin (mg/L), cytogenetic abnormalities as determined by fluorescence in situ hybridization (FISH), thrombocyte counts, albumin, and LDH. These prognostic factors will be determined at baseline, before the first daratumumab infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Niels W van de Donk, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] van de Donk NW, Janmaat ML, Mutis T, Lammerts van Bueren JJ, Ahmadi T, Sasser AK, Lokhorst HM, Parren PW. Monoclonal antibodies targeting CD38 in hematological malignancies and beyond. Immunol Rev. 2016 Mar;270(1):95-112. doi: 10.1111/imr.12389. PMID 26864107
- [Result] Lokhorst HM, Plesner T, Laubach JP, Nahi H, Gimsing P, Hansson M, Minnema MC, Lassen U, Krejcik J, Palumbo A, van de Donk NW, Ahmadi T, Khan I, Uhlar CM, Wang J, Sasser AK, Losic N, Lisby S, Basse L, Brun N, Richardson PG. Targeting CD38 with Daratumumab Monotherapy in Multiple Myeloma. N Engl J Med. 2015 Sep 24;373(13):1207-19. doi: 10.1056/NEJMoa1506348. Epub 2015 Aug 26. PMID 26308596
- [Result] Nijhof IS, Groen RW, Lokhorst HM, van Kessel B, Bloem AC, van Velzen J, de Jong-Korlaar R, Yuan H, Noort WA, Klein SK, Martens AC, Doshi P, Sasser K, Mutis T, van de Donk NW. Upregulation of CD38 expression on multiple myeloma cells by all-trans retinoic acid improves the efficacy of daratumumab. Leukemia. 2015 Oct;29(10):2039-49. doi: 10.1038/leu.2015.123. Epub 2015 May 15. PMID 25975191
- [Derived] Frerichs KA, Minnema MC, Levin MD, Broijl A, Bos GMJ, Kersten MJ, Mutis T, Verkleij CPM, Nijhof IS, Maas-Bosman PWC, Klein SK, Zweegman S, Sonneveld P, van de Donk NWCJ. Efficacy and safety of daratumumab combined with all-trans retinoic acid in relapsed/refractory multiple myeloma. Blood Adv. 2021 Dec 14;5(23):5128-5139. doi: 10.1182/bloodadvances.2021005220. PMID 34625791